CLINICAL TRIAL: NCT07247162
Title: A Double-blind, Randomised, 30-week Placebo-controlled Phase IV Study to Assess the Efficacy and Safety of Osilodrostat in Patients With Hypertension Caused by Hypercortisolaemia Due to Cushing's Syndrome
Brief Title: Osilodrostat in Patients With Hypertension Caused by Hypercortisolaemia Due to Cushing's Syndrome
Acronym: LINC CARE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCI699-RECAG-CL-0615; 2025-524649-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Hypercortisolemia; Cushing Syndrome
Keywords: osilodrostat; hypertension; hypercolesterolaemia; cushing's syndrome
MeSH Terms: conditions — Hypertension; ACTH Syndrome, Ectopic; Cushing Syndrome | interventions — Osilodrostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCI699 (osilodrostat) (Experimental): 1 mg QOD
  Interventions: Drug: Osilodrostat
- Placebo (Experimental): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Osilodrostat — Osilodrostat tablets 1 mg and 5 mg for oral useOsilodrostat tablets 1 mg and 5 mg for oral use.During the 18-week titration phase, the dose of the medication will be titrated every 3 weeks based on the cortisolaemic and clinical response to treatment. An independent endocrinologist titration committee will be applied to provide recommendations on dose-titration based on biochemical and clinical response. At the end of the 18-week dose titration phase, participants will enter a 12-week dose maintenance phase, which is also blinded. They will continue with the dose they were receiving at the end of the dose titration phase, unless there is a need to down-titrate or to stop the study medication for safety purposes.
  Arms: LCI699 (osilodrostat)
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
Osilodrostat has proven to be a safe and efficacious treatment for patients with CS. Demonstrating normalisation of hypercortisolaemia and in patients with hypertension and/or dysglycaemia clinically relevant and statistically significant reductions in blood pressure and glycaemia. This study aims at providing additional evidence on the safety, efficacy and appropriate dosing of osilodrostat in patients with CS, who have hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Able to provide and have provided signed written informed consent prior to study participation
3. Diagnosis of endogenous Cushing's Syndrome
4. mUFC values from two 24h urinary collections > ULN and ≤ 2x ULN
5. Participants with uncontrolled hypertension on stable doses of BP lowering medications (for at least 4 weeks); qualifying BP measurements by ABPM taken prior to randomisation defined as: Average of 24h ABPM SBP ≥ 135 or DBP ≥ 85 mmHg
6. Participants under glucocorticoid replacement therapy can be recruited only if this therapy has been already stopped for at least seven days or 5 half-lives prior to screening, whichever was longer
7. Not taking any drug therapy for CS. The following minimum periods without these medications need to be completed before baseline assessments:

   1. Steroidogenesis inhibitors (e.g. ketoconazole, metyrapone): 1 week
   2. Mifepristone: 3 weeks
   3. SC Pasireotide: 1 week
   4. Pasireotide LAR: 3 months
   5. Cabergoline: 4 weeks
8. Able to take oral medication and be willing to comply with the requirements of the study

Exclusion Criteria:

1. Previously treated with osilodrostat less than 12 weeks prior to start of screening
2. Known hypersensitivity to osilodrostat
3. Presence of any severe and/or uncontrolled medical condition or other conditions that could affect participation in the study
4. Participants who are scheduled for a surgery to treat CS within 32 weeks of randomisation to the study drug
5. Presence of a known "long term" history of both hypertension and diabetes (defined as both hypertension and diabetes diagnosed >10 years prior to the initial diagnosis of endogenous CS)
6. History of cyclic Cushing's Syndrome with fluctuating clinical manifestations
7. Participants with pseudo-CS
8. Participants with compression of the optic chiasm due to a macroadenoma or participants at high risk of compression of the optic chiasm (tumour within 2 mm of optic chiasm)
9. Pituitary radiation therapy within 3 years of screening
10. Ectopic ACTH syndrome or adrenocortical carcinoma with a life expectancy of <3 years or receiving chemotherapy
11. Having received prior mitotane treatment
12. Participants who are shift workers or have conditions that can affect the measurement of late night salivary cortisol (LNSC) or the LDDST
13. Poorly controlled diabetes mellitus with a baseline HbA1c > 10.5%
14. Poorly controlled BP defined as: Average SBP ≥ 170 or average DBP ≥ 110 mmHg as measured by the 24h ABPM
15. Participants who are hypothyroid and not on adequate replacement therapy
16. History of major surgery/surgical therapy for any cause within 1 month before entering the study.
17. Presence of bradycardia and/or QT-related exclusion criteria
18. Total bilirubin > 1.5 x ULN and ALT or AST > 3 x ULN
19. Participation in any clinical investigation within 4 weeks prior to screening or longer if required by local regulation (Use of an investigational drug within 1 month prior to dosing)
20. Occurrence of any significant acute illness within the three weeks prior to dosing/randomisation
21. Female participants who are pregnant, intending to become pregnant or breastfeed during the study or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
22. Women of childbearing potential (WOCBP) who are unwilling to use highly effective contraception methods
23. Potentially unreliable or vulnerable participants (e.g. person kept in detention) and those judged by the Investigator to be unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of osilodrostat on the proportion of participants with normalisation of urinary-free cortisol (UFC) | 30 weeks
  Proportion of participants with normalisation of the 24h-mUFC (as measured by the mean of the UFC concentrations of two 24-h urine collections ≤1xULN)